CLINICAL TRIAL: NCT04365244
Title: Pruritus and Melanoma and Cutaneous Carcinomas Treated With Immunotherapy (PRURICHECKPOINT)
Brief Title: Pruritus and Melanoma and Cutaneous Carcinomas Treated With Immunotherapy
Acronym: PRURICHECKPOIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PRURICHECKPOIN
Record Dates: First submitted 2020-04-16; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2019-04

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune checkpoint inhibitors (ICIs) are commonly used in the therapeutic arsenal of metastatic melanoma, Merkel cell carcinoma and cutaneous squamous cell carcinoma, thanks to their inhibiting effects on cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA4) and anti-programmed death-1 (anti-PD1) respectively. These treatments can induce numerous cutaneous and non-cutaneous adverse effects that are mainly due to their immunological action. Their most frequent adverse effects are dysthyroidism, autoimmune hepatitis, colitis and skin disorders. Among those, pruritus is frequently reported as a side effect of these treatments. Its incidence has been estimated between 11% and 47%. Pruritus can deeply affect the patient's quality of life and may lead to treatment discontinuation. Until now, ICI-related pruritus has been poorly studied and it is not understood. In the literature, data on the presence and characteristics of pruritus in patients treated by ICIs were provided, without analyzing the causes of this pruritus. Indeed, it is not known if the occurrence of pruritus is related to direct or indirect effects of ICIs. Some authors reported a correlation between the occurrence of cutaneous adverse events under ICIs and the survival. The principal aim of our study was to analyze the putative causes of pruritus occurring in patients treated with ICIs for melanomas and cutaneous carcinomas. The other objectives were to assess the association between the occurrence of pruritus and survival, and between the other adverse events and pruritus.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older,
* treated with ICIs (nivolumab, pembrolizumab, ipilimumab, cemiplimab) for melanoma, squamous cell carcinoma or Merkel cell carcinoma
* not having formulated any opposition

Exclusion Criteria:

* age under 18 years,
* adults not legally competent,
* presence of pruritus at the inclusion,
* participation refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with ICIs (nivolumab, pembrolizumab, ipilimumab or cemiplimab)
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
putative causes of pruritus | through study completion, an average of 1 year
  questionnaire

SECONDARY OUTCOMES:
presence of other side effects | through study completion, an average of 1 year
  questionnaire
survival | through study completion, an average of 1 year
  questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - CH de Landerneau, Landerneau

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning six month and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.